CLINICAL TRIAL: NCT01392703
Title: Open-label, Randomized, 3-period, 3-treatment Crossover, Bioequivalence Study Comparing Dasatinib (BMS-354825) Liquid Formulation and the Dispersed Tablet Formulation Relative to the Reference Tablet Formulation in Health Subjects
Brief Title: Pharmacokinetic Study Comparing Blood Levels of Dasatinib in Healthy Participants Who Received the Tablet Formulation With Those Who Received Liquid and Tablet-dispersed Formulations
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: CA180-352
Record Dates: First submitted 2011-07-11; First posted 2011-07-12 (Estimated); Results first posted 2013-02-11 (Estimated); Last update posted 2013-02-11 (Estimated); Status verified 2013-01

CONDITIONS: Pharmacokinetic Study in Healthy Participants
MeSH Terms: interventions — Dasatinib; Tablets; Fluid Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Dasatinib, 100 mg as tablets + water (Other): Treatment A. Participants were randomized to and received treatment in 1 of 6 sequences (ABC, ACB, BCA, BAC, CAB, or CBA), administered over 3 1-day treatment periods (Days 1, 5, and 9), with treatment changing to next in the sequence at start of each new period. A 3-day washout period followed treatment periods 1 and 2.
  Interventions: Drug: Dasatinib as tablets
- Dasatinib, 100 mg as liquid + water (Other): Treatment B. Participants were randomized to and received treatment in 1 of 6 sequences (ABC, ACB, BCA, BAC, CAB, or CBA), administered over 3 1-day treatment periods (Days 1, 5, and 9), with treatment changing to next in the sequence at start of each new period. A 3-day washout period followed treatment periods 1 and 2.
  Interventions: Drug: Dasatinib as liquid
- Dasatinib, 100 mg as tablets in orange juice + water (Other): Treatment C. Participants were randomized to and received treatment in 1 of 6 sequences (ABC, ACB, BCA, BAC, CAB, or CBA), administered over 3 1-day treatment periods (Days 1, 5, and 9), with treatment changing to next in the sequence at start of each new period. A 3-day washout period followed treatment periods 1 and 2.
  Interventions: Drug: Dasatinib as dispersed tablets

INTERVENTIONS:
Drug: Dasatinib as tablets — 2 50-mg tablets plus 240 mL noncarbonated, nonrefrigerated water. Oral, single dose, 1 day
  Other Names: Dasatinib/BMS-354825
  Arms: Dasatinib, 100 mg as tablets + water
Drug: Dasatinib as liquid — 100 mg administered as 10 mL of liquid drug (10 mg/mL) plus 230 mL noncarbonated, nonrefrigerated water. Oral, single dose, 1 day
  Other Names: Dasatinib/BMS-354825
  Arms: Dasatinib, 100 mg as liquid + water
Drug: Dasatinib as dispersed tablets — 2 50-mg dispersed tablets in 30 mL of 100% orange juice followed by 15 mL of orange juice plus 195 mL noncarbonated, nonrefrigerated water. Liquid (oral solution), single dose, 1 day.
  Other Names: Dasatinib/BMS-354825
  Arms: Dasatinib, 100 mg as tablets in orange juice + water

SUMMARY:
The purpose of the study is to compare the blood levels of dasatinib in healthy participants who received tablet formulation with those of healthy participants who received liquid and tablet-dispersed formulations of the drug.

ELIGIBILITY:
Key Inclusion Criteria:

* Healthy participants, defined as having no clinically relevant deviation from normal in medical history, physical examination, electrocardiogram (ECG) findings, and clinical laboratory tests findings.
* Body mass index of 18 to 32 kg/m^2, inclusive
* Age from 18 to 55 years
* Men and women who were not of childbearing potential (ie, who were postmenopausal or surgically sterile)
* All women must have had a negative serum or urine pregnancy test result(minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin) at screening and within 24 hours prior to dosing with study drug
* Women must not have been breastfeeding
* Sexually active fertile men with female partners of childbearing potential were required to abide by the requirement to use effective birth control for the entire study and for 90 days after the date of last treatment
* Men must have agreed not to donate sperm for the entire study and for 90 days after the day of last study treatment
* Participants must have agreed not to make blood donations, including red blood cells, plasma, platelets, or whole blood, for the entire study and for 8 weeks after the day of last study treatment

Key Exclusion Criteria:

* Any significant acute or chronic medical illness
* Current or recent (within 3 months of study drug administration) disease of the gastrointestinal (GI) tract that may impact drug absorption and may affect pharmacokinetics of the study drugs or any GI tract surgery that may impact drug absorption
* Any major surgery, as determined by the investigator, within 4 weeks of dosing in Period 1
* Blood transfusion within 4 weeks of study drug administration
* Donation of >400 mL of blood within 8 weeks prior to study dosing or donation of plasma within 4 weeks prior to study dosing
* Inability to tolerate oral medication
* Inability to tolerate orange juice
* Inability to undergo venipuncture and/or tolerate venous access
* Use of tobacco or nicotine-containing products within 6 months prior to check-in, or positive nicotine test at screening and/or check-in
* Consumption of more than 3 cups of coffee or other caffeine-containing products a day, or 5 cups of tea a day
* Recent (within 6 months of study drug administration) drug or alcohol abuse
* Positive blood screen for hepatitis C antibody; hepatitis B surface antigen; and HIV-1, HIV-2, or HIV antibody
* History of any significant drug allergy or asthma
* Evidence of organ dysfunction or any clinically relevant deviation from normal in physical examination, ECG findings, vital signs, or clinical laboratory test findings.
* Any of the following on 12-lead ECG prior to study drug administration, confirmed by repeat ECG:

  * PR ≥210 ms
  * QRS ≥120 ms
  * QT ≥500 ms
  * QTcF ≥450 ms

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 141 (Actual)
Dates: Start 2011-07; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Healthcare Discoveries Inc., San Antonio, Texas, United States

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 141 participants were enrolled, of which 78 were randomized to and received treatment in 1 of 6 sequences(ABC, ACB, BCA, BAC, CAB, or CBA), administered over 3 1-day treatment periods (Days 1, 5, and 9), with treatment changing to next in the sequence at start of each new period. A 3-day washout period followed treatment periods 1 and 2.
Groups:
- Dasatinib, 100 mg as Tablets + Water: Treatment A: Participants received a single oral dose of dasatinib, 100 mg, administered as 2 50-mg tablets, plus 240 mL of noncarbonated, nonrefrigerated water. All doses were administered in the fasted state. A 3-day washout period followed the treatment period.
- Dasatinib, 100 mg as Liquid + Water: Treatment B: Participants received a single oral dose of dasatinib, 100 mg, administered as 10 mL of reconstituted suspension of dasatinib powder for oral suspension (10 mg dasatinib/mL) with 230 mL of noncarbonated, nonrefrigerated water. All doses were administered in the fasted state. A 3-day washout period followed the treatment period.
- Dasatinib, 100 mg as Tablets in Orange Juice + Water: Treatment C: Participants received a single oral dose of dasatinib, 100 mg, administered as 2 50-mg tablets dispersed in 30 mL of 100% orange juice, followed by 15 mL of orange juice as a rinsing solution plus 195 mL noncarbonated, nonrefrigerated water. All doses were administered in the fasted state.
Period: Day 1
Arm/Group | Dasatinib, 100 mg as Tablets + Water | Dasatinib, 100 mg as Liquid + Water | Dasatinib, 100 mg as Tablets in Orange Juice + Water
Started | 26 | 26 | 26
Completed | 26 | 26 | 26
Not Completed | 0 | 0 | 0
Period: Day 5
Arm/Group | Dasatinib, 100 mg as Tablets + Water | Dasatinib, 100 mg as Liquid + Water | Dasatinib, 100 mg as Tablets in Orange Juice + Water
Started | 26 | 25 (1 participant no longer met dosing criteria and dropped out during washout period prior to Day 5.) | 26
Completed | 26 | 25 | 26
Not Completed | 0 | 0 | 0
Period: Day 9
Arm/Group | Dasatinib, 100 mg as Tablets + Water | Dasatinib, 100 mg as Liquid + Water | Dasatinib, 100 mg as Tablets in Orange Juice + Water
Started | 26 | 26 | 25
Completed | 26 | 26 | 25
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Treated
Number analyzed (Participants) | 78
Age Continuous [Mean (Standard Deviation); unit: years] | 36.5 (8.75)
Age, Customized [Number; unit: Participants]
  Younger than 65 years | 78
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 71
Race/Ethnicity, Customized [Number; unit: Participants]
  Hispanic/Latino | 39
  Not Hispanic/Latino | 39

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Concentration (Cmax) of Dasatinib
Description: Single-dose pharmacokinetic parameters, including Cmax, were derived using noncompartmental methods from plasma dasatinib concentration-time data.
Time Frame: Days 1-2, Days 5-6, and Days 9-10
Population: All participants who received at least 1 dose of any study drug and had pharmacokinetic data available.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Dasatinib, 100 mg as Tablets + Water | Dasatinib, 100 mg as Liquid + Water | Dasatinib, 100 mg as Tablets in Orange Juice + Water
Number analyzed (Participants) | 78 | 77 | 77
ng/mL | 114 (51) | 106 (53) | 110 (50)

2. Primary Outcome: Area Under the Plasma Concentration-time Curve From Zero to the Last Time of the Last Quantifiable Concentration (AUC[0-T])of Dasatinib
Description: Single-dose pharmacokinetic, such as AUC(0-T),parameters were derived using noncompartmental methods from plasma dasatinib concentration-time data.
Time Frame: Days 1-2, Days 5-6, and Days 9-10
Population: All participants who received at least 1 dose of any study drug and had pharmacokinetic data available.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Dasatinib, 100 mg as Tablets + Water | Dasatinib, 100 mg as Liquid + Water | Dasatinib, 100 mg as Tablets in Orange Juice + Water
Number analyzed (Participants) | 78 | 77 | 77
ng*h/mL | 374 (45) | 327 (44) | 342 (42)

3. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero Extrapolated to Infinity (AUC[0-INF]) of Dasatinib
Description: Single-dose pharmacokinetic parameters, such as AUC(0-INF) were derived using noncompartmental methods from plasma dasatinib concentration-time data.
Time Frame: Days 1-2, Days 5-6, and Days 9-10
Population: All participants who received at least 1 dose of any study drug and had pharmacokinetic data available.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Dasatinib, 100 mg as Tablets + Water | Dasatinib, 100 mg as Liquid + Water | Dasatinib, 100 mg as Tablets in Orange Juice + Water
Number analyzed (Participants) | 75 | 77 | 77
ng*h/mL | 429 (39) | 338 (43) | 353 (41)

4. Secondary Outcome: Time of Maximum Observed Plasma Concentration (Tmax) of Dasatinib
Description: Single-dose pharmacokinetic parameters, such as Tmax, were derived using noncompartmental methods from plasma dasatinib concentration-time data.
Time Frame: Days 1-2, Days 5-6, and Days 9-10
Population: All participants who received at least 1 dose of any study drug and had pharmacokinetic data available.
Measure: Median (Full Range); unit: Hours
Arm/Group | Dasatinib, 100 mg as Tablets + Water | Dasatinib, 100 mg as Liquid + Water | Dasatinib, 100 mg as Tablets in Orange Juice + Water
Number analyzed (Participants) | 78 | 77 | 77
Hours | 1.00 [0.25 to 3.00] | 0.53 [0.50 to 3.00] | 0.50 [0.50 to 4.00]

5. Secondary Outcome: Half-life of Dasatinib
Time Frame: Days 1-2, Days 5-6, and Days 9-10
Population: All participants who received at least 1 dose of any study drug and had pharmacokinetic data available.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Dasatinib, 100 mg as Tablets + Water | Dasatinib, 100 mg as Liquid + Water | Dasatinib, 100 mg as Tablets in Orange Juice + Water
Number analyzed (Participants) | 75 | 77 | 77
Hours | 4.96 (1.31) | 4.82 (1.17) | 4.91 (1.25)

6. Secondary Outcome: Number of Participants With at Least 1 Adverse Event (AE), With at Least 1 Treatment-related AE, Who Discontinued Due to AEs, and With at Least 1 Serious Adverse Event (SAE)
Description: An AE is any new untoward medical occurrence or worsening of a preexisting medical condition in a patient or clinical investigation participant who has received an investigational (medicinal) product that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of investigational product, whether or not considered related to the investigational product. An SAE is an untoward medical event that at any dose results in death, persistent or significant disability/incapacity; is life-threatening or a congenital anomaly/birth defect; or requires or prolongs hospitalization; is an important medical event that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the participant or may require medical or surgical intervention.
Time Frame: Continually from enrollment through Day 9 and at study discharge on Day 10
Population: All participants who received at least 1 dose of any study drug.
Measure: Number; unit: Participants
Arm/Group | Dasatinib, 100 mg as Tablets + Water | Dasatinib, 100 mg as Liquid + Water | Dasatinib, 100 mg as Tablets in Orange Juice + Water
Number analyzed (Participants) | 78 | 77 | 77
Participants
  At least 1 AE | 42 | 44 | 35
  At least 1 treatment-related AE | 39 | 43 | 34
  Discontinuation due to AEs | 0 | 0 | 0
  At least 1 SAE | 0 | 0 | 0

7. Secondary Outcome: Number of Participants With Clinically Significant Changes in Vital Signs or Electrocardiogram (ECG) Findings
Description: Blood pressure and heart rate were measured after the participant had been seated quietly for at least 5 minutes. ECG findings were recorded after the participant had been supine for at least 5 minutes. Clinically significant as reported by principal investigator.
Time Frame: Day -1, Screening, and Days 1, 5, 9 and 10 (at study discharge)
Population: All participants who received at least 1 dose of any study drug.
Measure: Number; unit: Participants
Arm/Group | All Treated
Number analyzed (Participants) | 78
Participants
  Respiratory rate | 0
  Temperature | 0
  Systolic blood pressure | 0
  Diastolic blood pressure | 0
  Heart rate | 0
  QT and QTc Intervals | 0
  QRS and PR intervals | 0

8. Secondary Outcome: Number of Participants With Marked Abnormalities in Results of Clinical Laboratory Tests
Description: Criteria for normal: bilirubin (0.2 to 1.3 mg/dL); lactate dehydrogenase (101 to 227 U/L); eosinophils (0.06 to 0.87*103 c/μL); erythrocytes (4.2 to 5.8*10^6 c/μL). Participants were required to fast for a minimum of 4 hours prior to the collection of specimens for clinical laboratory tests at screening and for at least 8 hours prior to collection on Day -1. Marked abnormalities were reported for the treatment regiment that participants received just prior to clinical laboratory testing.
Time Frame: Day -1, Screening, and Day 9 of current treatment regimen
Population: All participants who received at least 1 dose of any study drug.
Measure: Number; unit: Participants
Arm/Group | Dasatinib, 100 mg as Tablets + Water | Dasatinib, 100 mg as Liquid + Water | Dasatinib, 100 mg as Tablets in Orange Juice + Water
Number analyzed (Participants) | 78 | 77 | 77
Participants
  Elevated bilirubin | 0 | 0 | 1
  Elevated lactate dehydrogenase | 0 | 1 | 0
  Blood in urine (2+) | 1 | 0 | 0
  Elevated eosinophils | 0 | 0 | 1
  Low erythrocytes | 1 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Dasatinib, 100 mg as Tablets + Water | Dasatinib, 100 mg as Liquid + Water | Dasatinib, 100 mg as Tablets in Orange Juice + Water
Serious Adverse Events (participants affected / at risk) | 0/78 | 0/77 | 0/77
Other Adverse Events (participants affected / at risk) | 42/78 | 44/77 | 35/77
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dasatinib, 100 mg as Tablets + Water (N=78) | Dasatinib, 100 mg as Liquid + Water (N=77) | Dasatinib, 100 mg as Tablets in Orange Juice + Water (N=77)
Nausea (Gastrointestinal disorders) | 2 | 1 | 4
Headache (Nervous system disorders) | 40 | 43 | 35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.